CLINICAL TRIAL: NCT07162012
Title: The Safety and Efficacy of Anti-EBV Autologous TCR-T Cell Injection for Treating Relapsed/Refractory EBV-positive Lymphoma Patients With HLA-A11:01
Brief Title: Safety and Efficacy of Anti-EBV Autologous TCR-T Cell Injection in Relapsed/Refractory EBV-Positive Lymphoma
Acronym: Anti-EBV TCR-T
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Director of Department of Hematology, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY-EBV-TCR-T-202505
Record Dates: First submitted 2025-08-31; First posted 2025-09-09 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: NK/T-cell Lymphoma; Peripheral T-cell Lymphoma (PTCL); DLBCL
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Intervention Model Description: Using a rapid titration combined with a "3+3" design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- EBV-TCR-T (Experimental)
  Interventions: Drug: EBV TCR-T

INTERVENTIONS:
Drug: EBV TCR-T — After signing the informed consent form and completing screening according to the inclusion/exclusion criteria, eligible subjects will be sequentially assigned to the following dose cohorts of TCR-T cells (single administration): 1×10⁶ TCR-T cells/kg, 2.5×10⁶ TCR-T cells/kg, 5×10⁶ TCR-T cells/kg, and 10×10⁶ TCR-T cells/kg.
  The first dose cohort (1×10⁶ TCR-T cells/kg) will use a rapid titration approach. If no significant safety issues occur within 28 days after infusion-defined as ≥Grade 3 non-hematologic toxicity, Grade 4 hematologic toxicity lasting more than 28 days (excluding disease- or chemotherapy-related causes), ≥Grade 2 neurotoxicity, or ≥Grade 3 cytokine release syndrome (CRS)-the next dose cohort will be initiated. If a dose-limiting toxicity (DLT) occurs, evaluation will be performed after 6 subjects have been treated.
  The subsequent three dose cohorts will follow a "3+3" dose-escalation design, with 3-6 subjects per cohort receiving a single infusion. For subjects in th

SUMMARY:
This study will test whether anti-EBV autologous TCR-T cell injection is safe and effective for patients with relapsed or refractory EBV-positive lymphoma who have HLA-A11:01. Researchers will look at safety, tolerability, and the maximum tolerated dose or recommended dose for future studies.

The study will also measure how the infused TCR-T cells expand and persist in the body, changes in EBV DNA levels and T-cell subgroups in the blood, and whether the treatment shows early signs of clinical benefit. Researchers will also explore whether the treatment causes an immune response against the infused cells.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years, male or female.
2. HLA genotype at locus A is 11:01.
3. Disease diagnosis and status:

   1. Histologically or cytologically confirmed EBV-positive lymphoma (tumor tissue must be EBER-positive as confirmed by in situ hybridization [ISH] or fluorescence in situ hybridization [FISH]), with peripheral blood EBV viral load >10³ copies/mL by quantitative real-time PCR.
   2. Disease types include but are not limited to:

      NK/T-cell lymphoma (NK/TCL); Peripheral T-cell lymphoma (PTCL); Other types.
   3. Definition of relapse: appearance of new lesions at the primary site or other sites after achieving complete remission (CR).
   4. Definition of refractory disease (meeting any of the following):

   No partial remission (PR) after ≥4 cycles of standard therapy; No complete remission (CR) after ≥6 cycles of therapy; Failure to achieve CR after autologous hematopoietic stem cell transplantation; If best response is progressive disease (PD) or treatment is discontinued due to PD, no minimum cycle requirement applies.
4. Prior treatment requirements:

   a) For relapsed/refractory PTCL or NK/TCL, patients must have received at least one prior line of systemic therapy. For relapsed/refractory NK/TCL, patients must have received an asparaginase-containing regimen (patients with stage I/II nasal NK/TCL according to the CA staging system must have also received radiotherapy).
5. Measurable disease: At least one measurable lesion according to the 2014 Lymphoma Response Evaluation Criteria:

   1. Nodal lesions: longest diameter >15 mm on contrast-enhanced CT, MRI, or PET-CT;
   2. Extranodal lesions: longest diameter >10 mm. For patients with bone-marrow-only involvement who have no measurable lesions on imaging, the presence of ≥5% lymphoma cells in bone marrow biopsy or flow cytometry can be considered an evaluable lesion.
6. Adequate organ function, defined as:

   1. Hematologic: absolute neutrophil count ≥1×10⁹/L; hemoglobin ≥70 g/L; platelet count ≥50×10⁹/L;
   2. Hepatic: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × the upper limit of normal (ULN), and total bilirubin (TBIL) ≤ 1.5 × ULN (except when liver function abnormalities are attributable to the underlying disease);
   3. Renal: serum creatinine ≤1.5× ULN;
   4. Cardiac: left ventricular ejection fraction (LVEF) ≥50%;
   5. Coagulation: fibrinogen ≥1.0 g/L; activated partial thromboplastin time (APTT) ≤1.5× ULN; prothrombin time (PT) ≤1.5× ULN.
7. Expected survival >3 months.
8. ECOG performance status <3.
9. Contraception requirements:

   1. No pregnancy planned during the treatment period;
   2. Women of childbearing potential must have a negative pregnancy test and agree to use effective contraception during the study and for 4 months after the end of treatment.
10. Willingness to participate in the study, ability to sign informed consent, comply with the study protocol, and availability of peripheral venous access for lymphocyte collection.

Exclusion Criteria:

Subjects meeting any of the following conditions will not be eligible for enrollment:

1. History of other malignancies, except for:

   1. Basal cell carcinoma of the skin;
   2. Squamous cell carcinoma of the skin;
   3. Superficial bladder cancer;
   4. Carcinoma in situ of the cervix;
   5. Gastrointestinal mucosal carcinoma in situ;
   6. Other malignancies considered acceptable by the investigator (must have received curative treatment with no recurrence within the past 5 years).
2. Recent anti-tumor therapy: less than 4 weeks since last anti-cancer therapy (radiotherapy, chemotherapy, targeted therapy, immunotherapy, or local therapy), or less than 2 weeks since palliative radiotherapy.
3. Pregnant or breastfeeding women.
4. Presence of severe medical conditions such as intracranial hypertension, impaired consciousness, respiratory failure, or disseminated intravascular coagulation (DIC).
5. Severe organ dysfunction, including:

   NYHA class IV cardiac function; Child-Pugh class C liver function; Creatinine clearance <60 mL/min (by Cockcroft-Gault formula); Baseline oxygen saturation <92%.
6. Known active infections or positive screening results for:

   1. Hepatitis B virus (HBV): HBsAg positive, or HBcAb positive with HBV-DNA above the detection limit of the study center;
   2. Hepatitis C virus (HCV): HCV antibody positive and HCV RNA ≥ upper limit of normal (ULN);
   3. Human immunodeficiency virus (HIV) or Treponema pallidum (syphilis) antibody positive;
   4. Active tuberculosis (TB) (must be excluded by chest X-ray, sputum test, and clinical symptoms) or history of active TB;
   5. Severe acute or chronic infections requiring systemic treatment.
7. Active central nervous system (CNS) disease (e.g., tumor metastasis, infection, demyelinating disease), including untreated lesions, progressive disease on imaging or symptoms requiring urgent intervention, or requiring high-dose immunosuppressive therapy for control.
8. Receiving systemic corticosteroid therapy prior to screening and judged by the investigator to require long-term systemic corticosteroid treatment during the study (excluding inhaled or topical use); or receiving systemic corticosteroid treatment within 72 hours before cell infusion (excluding inhaled or topical use).
9. Presence of graft-versus-host disease (GVHD), defined as grade ≥2 acute GVHD or moderate/severe chronic GVHD, or current use of immunosuppressive therapy.
10. History of severe allergic reactions to drugs or excipients required in this study, or history of allergy to tocilizumab.
11. Any condition that, in the opinion of the investigator, makes the subject unsuitable for study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | treatment cycle (Day 1 to Day 28)
  To evaluate the incidence of dose-limiting toxicities (DLTs) of anti-EBV TCR-T cell injection in subjects with relapsed/refractory EBV-positive HLA-A11:01 lymphoma.
Maximum Tolerated Dose (MTD) | From Day 1 of treatment until the end of the dose-escalation phase
  Determination of the maximum tolerated dose of anti-EBV TCR-T cell injection.
Recommended Phase 2 Dose (RP2D) | At the completion of the dose-escalation phase
  Determination of the recommended dose for the expansion study based on safety, tolerability, and MTD.

SECONDARY OUTCOMES:
Expansion and persistence of EBV TCR-T cells | From Day 1 of infusion up to 24 months
  To evaluate the in vivo expansion and persistence of anti-EBV TCR-T cells after infusion
EBV DNA copies in peripheral blood | From Day 1 of infusion up to 24 months
  To evaluate the EBV DNA copy number in peripheral blood after infusion of anti-EBV TCR-T cells.
Changes in T-cell subsets in peripheral blood | From Day 1 of infusion up to 24 months
  To evaluate the changes in peripheral blood T-cell subsets after infusion of anti-EBV TCR-T cells.
Objective Response Rate (ORR) | At 3 months and 6 months after infusion
  Proportion of subjects achieving complete response (CR) or partial response (PR) following treatment with anti-EBV TCR-T cells.
Duration of Response (DOR) | From the first documented response (CR or PR) until disease progression/relapse or death, up to 24 months
  Duration of response in subjects with relapsed/refractory EBV-positive lymphoma treated with anti-EBV TCR-T cells.
Progression-Free Survival (PFS) | From infusion until documented disease progression or death, up to 24 months
  Progression-free survival following anti-EBV TCR-T cell treatment.
Overall Survival (OS) | From infusion until death from any cause, up to 24 months
  Overall survival following anti-EBV TCR-T cell treatment.

OTHER OUTCOMES:
Pharmacokinetic (PK) parameters | From Day 1 to Day 28 after infusion
  Maximum concentration (Cmax), time to maximum concentration (Tmax), and area under the curve (AUC0-28d) of anti-EBV TCR-T cells in peripheral blood.
Pharmacodynamic (PD) parameters | From Day 1 of infusion up to 24 months
  plasma cytokine levels at multiple time points after infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chou CC, Tsao CF, Liao CK, You HL, Wang MC, Huang WT. Analysis of latent T-cell epitopes in Epstein-Barr virus isolated from extranodal nasal-type natural killer/T-cell lymphoma in Taiwanese population. Exp Mol Pathol. 2021 Feb;118:104577. doi: 10.1016/j.yexmp.2020.104577. Epub 2020 Nov 23. PMID 33242451
- [Result] Barros MHM, Alves PDS. Contribution of the Epstein-Barr virus to the oncogenesis of mature T-cell lymphoproliferative neoplasms. Front Oncol. 2023 Sep 14;13:1240359. doi: 10.3389/fonc.2023.1240359. eCollection 2023. PMID 37781191
- [Result] Hinrichs CS, Restifo NP. Reassessing target antigens for adoptive T-cell therapy. Nat Biotechnol. 2013 Nov;31(11):999-1008. doi: 10.1038/nbt.2725. Epub 2013 Oct 20. PMID 24142051
- [Result] Heslop HE, Slobod KS, Pule MA, Hale GA, Rousseau A, Smith CA, Bollard CM, Liu H, Wu MF, Rochester RJ, Amrolia PJ, Hurwitz JL, Brenner MK, Rooney CM. Long-term outcome of EBV-specific T-cell infusions to prevent or treat EBV-related lymphoproliferative disease in transplant recipients. Blood. 2010 Feb 4;115(5):925-35. doi: 10.1182/blood-2009-08-239186. Epub 2009 Oct 30. PMID 19880495
- [Result] Okamoto A, Yanada M, Miura H, Inaguma Y, Tokuda M, Morishima S, Kanie T, Yamamoto Y, Mizuta S, Akatsuka Y, Yoshikawa T, Mizoguchi Y, Nakamura S, Okamoto M, Emi N. Prognostic significance of Epstein-Barr virus DNA detection in pretreatment serum in diffuse large B-cell lymphoma. Cancer Sci. 2015 Nov;106(11):1576-81. doi: 10.1111/cas.12812. Epub 2015 Oct 7. PMID 26353084
- [Result] Gao X, Li J, Wang Y, Liu S, Yue B. Clinical characteristics and prognostic significance of EBER positivity in diffuse large B-cell lymphoma: A meta-analysis. PLoS One. 2018 Jun 19;13(6):e0199398. doi: 10.1371/journal.pone.0199398. eCollection 2018. PMID 29920566
- [Result] Lu TX, Liang JH, Miao Y, Fan L, Wang L, Qu XY, Cao L, Gong QX, Wang Z, Zhang ZH, Xu W, Li JY. Epstein-Barr virus positive diffuse large B-cell lymphoma predict poor outcome, regardless of the age. Sci Rep. 2015 Jul 23;5:12168. doi: 10.1038/srep12168. PMID 26202875
- [Result] Song CG, Huang JJ, Li YJ, Xia Y, Wang Y, Bi XW, Jiang WQ, Huang HQ, Lin TY, Li ZM. Epstein-Barr Virus-Positive Diffuse Large B-Cell Lymphoma in the Elderly: A Matched Case-Control Analysis. PLoS One. 2015 Jul 29;10(7):e0133973. doi: 10.1371/journal.pone.0133973. eCollection 2015. PMID 26222726
- [Result] Ok CY, Papathomas TG, Medeiros LJ, Young KH. EBV-positive diffuse large B-cell lymphoma of the elderly. Blood. 2013 Jul 18;122(3):328-40. doi: 10.1182/blood-2013-03-489708. Epub 2013 May 6. PMID 23649469
- [Result] Healy JA, Dave SS. The Role of EBV in the Pathogenesis of Diffuse Large B Cell Lymphoma. Curr Top Microbiol Immunol. 2015;390(Pt 1):315-37. doi: 10.1007/978-3-319-22822-8_13. PMID 26424652
- [Result] Lesokhin AM, Ansell SM, Armand P, Scott EC, Halwani A, Gutierrez M, Millenson MM, Cohen AD, Schuster SJ, Lebovic D, Dhodapkar M, Avigan D, Chapuy B, Ligon AH, Freeman GJ, Rodig SJ, Cattry D, Zhu L, Grosso JF, Bradley Garelik MB, Shipp MA, Borrello I, Timmerman J. Nivolumab in Patients With Relapsed or Refractory Hematologic Malignancy: Preliminary Results of a Phase Ib Study. J Clin Oncol. 2016 Aug 10;34(23):2698-704. doi: 10.1200/JCO.2015.65.9789. Epub 2016 Jun 6. PMID 27269947
- [Result] Lim SH, Hong JY, Lim ST, Hong H, Arnoud J, Zhao W, Yoon DH, Tang T, Cho J, Park S, Ko YH, Kim SJ, Suh C, Lin T, Kim WS. Beyond first-line non-anthracycline-based chemotherapy for extranodal NK/T-cell lymphoma: clinical outcome and current perspectives on salvage therapy for patients after first relapse and progression of disease. Ann Oncol. 2017 Sep 1;28(9):2199-2205. doi: 10.1093/annonc/mdx316. PMID 28911074
- [Result] Grogg KL, Miller RF, Dogan A. HIV infection and lymphoma. J Clin Pathol. 2007 Dec;60(12):1365-72. doi: 10.1136/jcp.2007.051953. PMID 18042692
- [Result] Fox CP, Haigh TA, Taylor GS, Long HM, Lee SP, Shannon-Lowe C, O'Connor S, Bollard CM, Iqbal J, Chan WC, Rickinson AB, Bell AI, Rowe M. A novel latent membrane 2 transcript expressed in Epstein-Barr virus-positive NK- and T-cell lymphoproliferative disease encodes a target for cellular immunotherapy. Blood. 2010 Nov 11;116(19):3695-704. doi: 10.1182/blood-2010-06-292268. Epub 2010 Jul 29. PMID 20671118
- [Result] Kuppers R, Engert A, Hansmann ML. Hodgkin lymphoma. J Clin Invest. 2012 Oct;122(10):3439-47. doi: 10.1172/JCI61245. Epub 2012 Oct 1. PMID 23023715